CLINICAL TRIAL: NCT07004504
Title: MEnstrual Cycle pHase ANd dIabeteS Management
Acronym: MECHANISM
Status: Completed | Type: Observational
Sponsor: DCB Research AG (Other)
Responsible Party: Sponsor
Other Study IDs: MECHANISM
Record Dates: First submitted 2025-02-27; First posted 2025-06-04 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Insulin sensitivity; Menstrual cycle; Diabetes management
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single Arm: The study cohort consists of women with type 1 diabetes (T1D) who use continuous glucose monitoring (CGM) and insulin pumps to manage their diabetes. Participants will anonymously upload their glucose and insulin delivery data, along with self-reported menstrual cycle information. The study focuses on analyzing variations in insulin requirements and glycemic control across menstrual cycle phases, without introducing any direct interventions.

SUMMARY:
This study examines how menstrual cycle phases affect glycemic control and insulin requirements in women with type 1 diabetes (T1D). It aims to analyze differences in insulin needs and glucose levels between follicular and luteal phases using data from the Tidepool Data Platform. Key parameters include mean glucose, Time in Range (TIR), and total insulin administration. Secondary objectives involve assessing phase-specific glucose fluctuations, aggregated differences, and insulin adjustment strategies. The study follows a decentralized, anonymous data collection approach with participants using CGMs and insulin pumps or smart pens. Statistical analysis includes linear mixed-effects modeling to compare glycemic variability across cycle phases. Findings aim to enhance our understanding of diabetes management during the menstrual cycle and potentially inform future treatment strategies.

ELIGIBILITY:
Inclusion criteria

People are eligible to participate in the study if they:

* are living with T1D;
* are willing to upload diabetes-related data to the Tidepool Data Platform;
* are using a continuous glucose monitoring (CGM) system;
* are using an insulin pump or a smart pen for most of their insulin delivery;
* are willing to track and share their menstrual cycle data;
* are 18 years old or older;
* give consent to share their anonymized data for research.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes adults (18+) living with type 1 diabetes (T1D) who use a continuous glucose monitoring (CGM) system and either an insulin pump or a smart pen for insulin delivery. Participants must be willing to upload diabetes-related data to the Tidepool Data Platform, track and share their menstrual cycle data, and provide consent for their anonymized data to be used in research.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2024-12-29 (Actual)

PRIMARY OUTCOMES:
Mean glucose | Between 1 and 12 months
  Mean daily glucose based on CGM data

SECONDARY OUTCOMES:
Time in range (TIR) | Between 1 and 12 months
  Mean daily TIR based on CGM data
Time above range (TAR) | Between 1 and 12 months
  Mean daily TAR based on CGM data
Time belwo range (TBR) | Between 1 and 12 months
  Mean daily TBR based on CGM data
Total daily insulin | Between 1 and 12 months
  Mean daily total insulin based on insulin pump data
Total basal insulin | Between 1 and 12 months
  Mean daily total basal insulin based on insulin pump data
Total bolus insulin | Between 1 and 12 months
  Mean daily total bolus insulin based on insulin pump data

CONTACTS AND LOCATIONS:
Overall Officials: Martina Rothenbühler, PhD, Principal Investigator — DCB Research AG
Locations (1):
- DCB Research AG, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schiavon M, Dalla Man C, Kudva YC, Basu A, Cobelli C. Quantitative estimation of insulin sensitivity in type 1 diabetic subjects wearing a sensor-augmented insulin pump. Diabetes Care. 2014;37(5):1216-23. doi: 10.2337/dc13-1120. Epub 2013 Dec 6. PMID 24319120